CLINICAL TRIAL: NCT03441867
Title: Neuroimaging Biomarker for Seizures
Acronym: NIBMSZS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Providence VA Medical Center (U.S. Federal Agency)
Collaborators: University of Alabama at Birmingham (Other); Rhode Island Hospital (Other); Birmingham, Alabama VA Medical Center (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency); Ocean State Research Institute, Inc. (Other); Brown University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Award Number W81XWH-17-1-0619
Record Dates: First submitted 2017-12-29; First posted 2018-02-22 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Seizure Disorder; Seizure Disorder, Post Traumatic; Traumatic Brain Injury; Non-Epileptic Seizure; Conversion Disorder; Magnetic Resonance Imaging; Head Injury; Epilepsy
Keywords: Cognitive Behavioral Therapy; Veterans; Quality of Life; Stress Disorders, Post-Traumatic; Convulsion, Non-Epileptic; civilians; healthy volunteers
MeSH Terms: conditions — Epilepsy; Epilepsy, Post-Traumatic; Brain Injuries, Traumatic; Seizures; Conversion Disorder; Craniocerebral Trauma; Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Masking Description: The neuroimaging analysis will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- (CBT-Sz) - PNES (Experimental): Participants with history of a head injury and confirmed Psychogenic Non-Epileptic Seizures will complete 2 brain fMRI scans along with 12 weeks of one hour CBT-Sz sessions by a trained therapist.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Seizures
- (CBT-Sz) - PTE (Experimental): Participants with history of a head injury and confirmed Post-Traumatic Epilepsy (PTE) will complete 2 brain fMRI scans along with 12 weeks of one hour CBT-Sz sessions by a trained therapist.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Seizures
- TBI Control (Active Comparator): Participants with TBI will complete 2 brain fMRI scans.
  Interventions: Other: Standard Medical Care
- Healthy Volunteer (Active Comparator): Healthy control volunteers will complete 2 brain fMRI scans.
  Interventions: Other: Standard Medical Care

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Seizures — CBT-informed psychotherapy for patients with PNES and PTE
  Other Names: Cognitive Behavioral Therapy (CBT-Sz); (CBT-Sz) - PNES; (CBT-Sz) - PTE
  Arms: (CBT-Sz) - PNES; (CBT-Sz) - PTE
Other: Standard Medical Care — Observational - standard medical care
  Other Names: Treatment as Usual
  Arms: Healthy Volunteer; TBI Control

SUMMARY:
This multi-site study will examine patients with epilepsy (ES) following head injury [i.e., posttraumatic epilepsy (PTE)] and posttraumatic psychogenic Non-epileptic seizures (PNES) and will compare them to patients with traumatic brain injury (TBI) who do not have seizures using functional neuroimaging.

DETAILED DESCRIPTION:
Numerous Veterans and civilians have seizures, which can be epileptic or nonepileptic in nature. Epileptic seizures are caused by abnormal brain cell firing. Nonepileptic seizures appear similar to epileptic seizures, but are associated with traumatic experiences and underlying psychological stressors. Both types of seizure are common and disabling, and many patients with seizures do not have adequate control resulting in loss of quality of life.

In this proposed 3-site study ( Providence, RI and Birmingham, AL), which are epilepsy centers with expertise both in epilepsy and psychogenic nonepileptic seizures (PNES), we will enroll 88 patients with video-EEG confirmed PNES and 88 with confirmed post-traumatic epilepsy (PTE) and will obtain functional neuroimaging before and after they receive a behavioral treatment - Cognitive Behavioral Therapy for Seizures. The functional neuroimaging studies in these patients will be compared to patients with traumatic brain injury without seizures to test the hypothesis that the faulty processing of emotions and stress in patients with PNES/PTE and abnormal brain connectivity have unique signals in patients with seizures compared to Veterans without seizures and that the neuroimaging signatures can be modified using behavioral intervention.

Impact: This grant application for the first study investigating mechanisms of PNES and PTE will provide increased understanding of neural circuitry in PTE and PNES, which can inform PTE and PNES treatments and could change clinical neurologic and psychiatric practice for PTE and PNES.

Participants will be recruited at the Providence VA Medical Center, Rhode Island Hospital, and University of Alabama, Birmingham (UAB).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for PNES, ES and TBI (w/o PNES or ES) participants

  * Individuals with history of documented TBI (any severity).
  * Males and Females ages 18-60 years .
  * Women of child bearing potential, if currently using appropriate contraception.

Inclusion criteria of PNES and ES participants.

* Diagnosed by video/EEG with lone PNES or by EEG with lone ES.
* Patients must have at least 1 PNES or 1 ES during the year prior to enrollment.

Exclusion Criteria:

* Exclusion Criteria of PNES, ES and TBI (w/o PNES or ES) participants

  * Current or past year self-injurious behavior.
  * Current suicidal intent (BDI suicide question 9 score of >1).
  * Current or past year psychosis.
  * Pending litigation or current application for long term disability.
  * Active substance or alcohol use disorder (dependence), per discretion of the investigators.
  * Serious illness requiring systemic treatment or hospitalization; the participant either completes therapy or is clinically stable on therapy, for at least 30 days prior to study entry.
  * Inability to fill out the self-report surveys.
  * Women who are or/are attempting to become pregnant during the study.
  * Ineligible or unwilling to complete MRI imaging.
  * Inability to document TBI.

Exclusion Criteria for PNES and ES participants

* Inability or unwillingness to participate in CBT and assigned homework.
* Currently enrolled in cognitive therapy aimed at PNES (Current CBT or other psychotherapy may be administered).
* Concurrent mixed ES/PNES or equivocal video/EEG findings in discerning between ES and PNES will not be enrolled.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-09-14 (Estimated)

PRIMARY OUTCOMES:
Number of Epileptic Seizures | Baseline, Weeks 1,2,3,4,5,6,7,8,9,10,11,12, 8 months post baseline, 12 months post baseline
  epileptic seizure frequency (ES), collected prospectively, using a daily seizure calendar
Number of Nonepileptic Seizures (NES) | Baseline, Weeks 1,2,3,4,5,6,7,8,9,10,11,12, 8 months post baseline, 12 months post baseline
  psychogenic nonepileptic seizure (NES) frequency, collected prospectively, using a daily seizure calendar
Structural and Functional Neuroimaging | Baseline and week 13
  Brain MRI scans

SECONDARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | Baseline, Weeks 1,2,3,4,5,6,7,8,9,10,11,12, 8 months post baseline, 12 months post baseline
  The BDI-II assesses depression severity from "0" (no Depression-related symptom) to "3" (severe) on each question. The highest possible score is "51", relating to the worst outcome.
Beck Anxiety Inventory (BAI) | Baseline, Weeks 6 and 10, 8 months post baseline, 12 months post baseline
  The BDI-II assesses anxiety severity from "0" (no Anxiety-related symptom) to "3" (severe) on each question.
Quality of Life in Epilepsy-31 (QOLIE-31) | Baseline, Weeks 6 and 10
  his is a 31-item self-report scale used in the seizure population to evaluate Quality of Life. The lowest possible score is 0 and the highest possible score is 100, reflecting a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: W. Curt LaFrance, Jr., MD, MPH, Principal Investigator — Providence VA Medical Center; Jerzy Szarflarski, MD, Principal Investigator — University of Alabama at Birmingham
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Rhode Island Hospital, Providence, Rhode Island
  - Providence VA Medical Center, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LaFrance WC Jr, Baird GL, Barry JJ, Blum AS, Frank Webb A, Keitner GI, Machan JT, Miller I, Szaflarski JP; NES Treatment Trial (NEST-T) Consortium. Multicenter pilot treatment trial for psychogenic nonepileptic seizures: a randomized clinical trial. JAMA Psychiatry. 2014 Sep;71(9):997-1005. doi: 10.1001/jamapsychiatry.2014.817. PMID 24989152
- [Background] Salinsky M, Spencer D, Boudreau E, Ferguson F. Psychogenic nonepileptic seizures in US veterans. Neurology. 2011 Sep 6;77(10):945-50. doi: 10.1212/WNL.0b013e31822cfc46. PMID 21893668
- [Background] LaFrance WC Jr, Friedman JH. Cognitive behavioral therapy for psychogenic movement disorder. Mov Disord. 2009 Sep 15;24(12):1856-7. doi: 10.1002/mds.22683. No abstract available. PMID 19562779
- [Background] LaFrance WC Jr, Keitner GI, Papandonatos GD, Blum AS, Machan JT, Ryan CE, Miller IW. Pilot pharmacologic randomized controlled trial for psychogenic nonepileptic seizures. Neurology. 2010 Sep 28;75(13):1166-73. doi: 10.1212/WNL.0b013e3181f4d5a9. Epub 2010 Aug 25. PMID 20739647
- [Background] Reiter JM, Andrews DJ. A neurobehavioral approach for treatment of complex partial epilepsy: efficacy. Seizure. 2000 Apr;9(3):198-203. doi: 10.1053/seiz.1999.0374. PMID 10775516
- [Background] Elsas SM, Gregory WL, White G, Navarro G, Salinsky MC, Andrews DJ. Aura interruption: the Andrews/Reiter behavioral intervention may reduce seizures and improve quality of life - a pilot trial. Epilepsy Behav. 2011 Dec;22(4):765-72. doi: 10.1016/j.yebeh.2011.09.030. Epub 2011 Nov 6. PMID 22056814
- [Background] Michaelis R, Schonfeld W, Elsas SM. Trigger self-control and seizure arrest in the Andrews/Reiter behavioral approach to epilepsy: a retrospective analysis of seizure frequency. Epilepsy Behav. 2012 Mar;23(3):266-71. doi: 10.1016/j.yebeh.2011.11.023. Epub 2012 Feb 15. PMID 22341960
- [Background] Allendorfer JB, Szaflarski JP. Physiologic and cortical response to acute psychosocial stress in left temporal lobe epilepsy: response to a biochemical evaluation. Epilepsy Behav. 2014 Dec;41:312-3. doi: 10.1016/j.yebeh.2014.08.018. Epub 2014 Oct 11. No abstract available. PMID 25306199
- [Background] Szaflarski JP, Ficker DM, Cahill WT, Privitera MD. Four-year incidence of psychogenic nonepileptic seizures in adults in hamilton county, OH. Neurology. 2000 Nov 28;55(10):1561-3. doi: 10.1212/wnl.55.10.1561. PMID 11094115
- [Background] LaFrance WC Jr, Syc S. Depression and symptoms affect quality of life in psychogenic nonepileptic seizures. Neurology. 2009 Aug 4;73(5):366-71. doi: 10.1212/WNL.0b013e3181b04c83. PMID 19652140
- [Background] Szaflarski JP, Hughes C, Szaflarski M, Ficker DM, Cahill WT, Li M, Privitera MD. Quality of life in psychogenic nonepileptic seizures. Epilepsia. 2003 Feb;44(2):236-42. doi: 10.1046/j.1528-1157.2003.35302.x. PMID 12558580
- [Background] Voon V, Brezing C, Gallea C, Ameli R, Roelofs K, LaFrance WC Jr, Hallett M. Emotional stimuli and motor conversion disorder. Brain. 2010 May;133(Pt 5):1526-36. doi: 10.1093/brain/awq054. Epub 2010 Apr 5. PMID 20371508
- [Derived] Van Patten R, Cotton E, Chan L, Altalib H, Tocco K, Gaston TE, Grayson LP, Martin A, Fry S, Goodman A, Allendorfer JB, Blum A, Szaflarski JP, LaFrance WC Jr. Neurobehavioral Therapy Is Associated With Improvements in Social Functioning in Patients With Functional Seizures and Traumatic Brain Injury. J Clin Psychol. 2026 Jan;82(1):84-96. doi: 10.1002/jclp.70047. Epub 2025 Sep 25. PMID 40996372

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT03441867/Prot_SAP_001.pdf